CLINICAL TRIAL: NCT02309554
Title: A Phase I Postcoital Testing Study of the SILCS Diaphragm Used With 3% Nonoxynol-9 Gel, ContraGel, or No Gel
Brief Title: Postcoital Testing Study of the SILCS Diaphragm Used With 3% N-9 Gel, ContraGel, or No Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: A13-126
Record Dates: First submitted 2014-07-14; First posted 2014-12-05 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Contraception
Keywords: Contraception; Post coital test; Vaginal; Diaphragm
MeSH Terms: interventions — Nonoxynol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SILCS Diaphragm alone (Active Comparator): Participants will complete a post-coital test cycle with SILCS diaphragm alone.
  Interventions: Other: SILCS diaphragm
- SILCS Diaphragm with 3% Nonoxynol-9 Gel (Active Comparator): Participants will complete a post-coital test cycle with SILCS diaphragm used with 3% nonoxynol-9 gel.
  Interventions: Other: SILCS diaphragm used with 3% Nonoxynol-9; Other: SILCS diaphragm
- SILCS Diarphragm with ContraGel (Experimental): Participants will complete a post-coital test cycle with SILCS diaphragm used with ContraGel.
  Interventions: Other: SILCS diaphragm used with ContraGel; Other: SILCS diaphragm

INTERVENTIONS:
Other: SILCS diaphragm used with ContraGel — SILCS Diaphragm (branded as CAYA countoured diaphragm) is a single-size vaginal barrier method of contraception used with each sex act, made of silicone membrane with a nylon spring. ContraGel is a clear, water soluble greaseless gel packed in a metal tube.
  Arms: SILCS Diarphragm with ContraGel
Other: SILCS diaphragm used with 3% Nonoxynol-9 — SILCS Diaphragm (branded as CAYA countoured diaphragm) is a single-size vaginal barrier method of contraception used with each sex act, made of silicone membrane with a nylon spring. 3% Nonoxynol-9 (branded as Gynol II) is clear, unscented water soluble greaseless gel packed in plastic tubes with a vaginal applicator.
  Arms: SILCS Diaphragm with 3% Nonoxynol-9 Gel
Other: SILCS diaphragm — SILCS Diaphragm (branded as CAYA countoured diaphragm) is a single-size vaginal barrier method of contraception used with each sex act, made of silicone membrane with a nylon spring

SUMMARY:
This post coital test study is a Phase I multi-center, randomized, crossover, non-significant risk device study to be carried out at two clinical sites/centers. The products to be tested are the SILCS diaphragm with 3% Nonoxynol-9 Gel (N-9) (spermicide), the SILCS diaphragm with ContraGel, and the SILCS diaphragm alone. Participants will be randomized to the order of product use, with a goal of 10 participants completing the study.

DETAILED DESCRIPTION:
Each participant will be seen in approximately nine visits, over a period of 6-8 months, and will be contacted approximately 7 days after the final visit. Volunteers will be consented at Visit 1 and undergo procedures to confirm they are eligible to continue in the study.

Each participant will undergo four postcoital test (PCT) cycles:

1. The first PCT cycle will be a baseline cycle, done without the use of any product, in order to demonstrate the participant's ability to undergo normal ovulatory events and to produce receptive, midcycle cervical mucus. The partner's ability to produce motile sperm capable of penetrating the cervical mucus is also evaluated in this cycle.
2. Test PCT cycles will be carried out during the subsequent menstrual cycles using either the SILCS diaphragm with 3% N-9, the SILCS diaphragm with ContraGel, or the SILCS diaphragm alone following a sequence of randomized treatment. Cycles may need to be repeated depending on the characteristics of the cervical mucus and the number of sperm found in the vaginal pool and endocervical specimens.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 years, inclusive
2. General good health, by volunteer history and per investigator judgment
3. History of regular menstrual cycles of 24-35 days (inclusive), by volunteer report
4. History of Pap smears and follow-up consistent with standard medical practice as outlined in the Study Manual or willing to undergo a Pap smear at Visit 1
5. Willing to abstain from intercourse and use of vaginal products as required in the protocol
6. Willing to use non-spermicidal, lubricated condoms from the first day of each menstrual cycle until 72 hours before expected midcycle
7. In a mutually monogamous relationship for at least the last four months with a male partner who: 7a. Is at least 18 years old; 7b. Has no known risk for STIs; 7c. Is willing and able to comply with protocol requirements including sexual activity/ abstinence and condom use requirements; and 7d. Can engage in vaginal intercourse with the participant, with and without condoms, as specified in protocol
8. Protected from pregnancy by female tubal sterilization
9. Vaginal and cervical anatomy that, in the opinion of the investigator, lends itself to easy genital tract sample collection
10. Willing to give voluntary consent, sign an informed consent form and comply with study procedures as required by the protocol

Exclusion Criteria:

1. History of hysterectomy
2. Vasectomy in male partner
3. Sterility or known history of sperm dysfunction in male partner
4. Currently pregnant or within two calendar months from the last pregnancy outcome. Note: If recently pregnant must have had at least two spontaneous menses since pregnancy outcome
5. Current use of any hormonal contraceptive or a copper IUD, or use of Depo-Provera in the last 120 days
6. Currently breastfeeding or having breastfed an infant in the last two months, or planning to breastfeed during the course of the study
7. Significant gynecological abnormalities (including abnormal vaginal bleeding or excessive vaginal discharge)
8. Device does not appropriately fit volunteer, as determined by clinician
9. Inability to insert, position, and/or remove study device, by clinician or volunteer
10. History of sensitivity/allergy to 3% N-9, latex, ingredients in ContraGel, or silicone, for either the volunteer or her male partner
11. In the last six months, either the volunteer or her male partner diagnosed with or treated for any STI or pelvic inflammatory disease. Note: Women with a history of genital herpes or condylomata who have been asymptomatic for at least six months may be considered for eligibility
12. Positive test for Trichomonas vaginalis, Neisseria gonorrhea or Chlamydia trachomatis
13. Deep epithelial genital findings such as abrasions, ulcerations, and lacerations, or vesicles suspicious for a sexually transmitted infection
14. Positive test for HIV
15. Chronic or acute vulvar or vaginal symptoms (pain, irritation, spotting, etc.)
16. Known current drug or alcohol abuse which could impact study compliance
17. Participation in any other investigational trial within the last 30 days or planned participation in any other investigational trial during the study
18. History of gynecological procedures (including genital piercing) on the external genitalia, vagina or cervix within the last 14 days
19. Abnormal finding on laboratory or physical examination or a social or medical condition in either the volunteer or her male partner which, in the opinion of the investigator, would make participation in the study unsafe or would complicate interpretation of data

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2014-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Proportion of women with an average of fewer than 5 progressively motile sperm per high powered field (HPF) as a measure of preliminary effectiveness | 2-3 hours following coitus
  Fewer than 5% progressively motile sperm per high power field is considered indicative of acceptable barrier function. Will be calculated separately for each test cycle.
Per-women average number (across 9 HPFs) of progressively motile sperm per HPF as a measure of preliminary effectiveness. | 2-3 hours following coitus
  Mean, median, standard deviation and IQR will be assessed for the baseline cycle and during each test PCT, across all women. Qualitative assessments of change from baseline, if any, will be based on medians and IQRs.

SECONDARY OUTCOMES:
Number of treatment emergent adverse experiences among female participants as a measure of safety | Beginning at Visit 2 through 7-10 days after the final study visit; an average of 6-8 months
  Urogenital, product-related, and/or serious AEs will be assessed
Number of treatment emergent adverse experiences among male partners as a measure of safety | Beginning at Visit 2 through 7-10 days after the final study visit; an average of 6-8 months
  Urogenital, product-related, and/or serious AEs will be assessed

CONTACTS AND LOCATIONS:
Locations (2):
- Clinical Research Center, Eastern Virginia Medical School, Norfolk, Virginia, United States
- ProFamilia, Santo Domingo, Dominican Republic